CLINICAL TRIAL: NCT04055662
Title: A Comparison of Post-Operative Analgesia Requirements In Recreational Cannabis Users
Brief Title: A Comparison of Post-Operative Analgesia Requirements In Recreational Cannabis Users Versus Cannabis Naïve Inflammatory Bowel Disease Patients
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 2108.2.7
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2019-08

CONDITIONS: Cannabis Use, Opioid Consumption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cannabis users
- Cannabis naive

SUMMARY:
Cannabis is a drug that is widely used for recreational purpose. In most patients undergoing surgery, opioids are the most widely used mode of pain relief, during and following surgery. Anecdotally it has been observed that cannabis users required unexpectedly high doses of opioids. The purpose of this study is to compare opioid requirements between cannabis users and non- users after the surgery. Currently, post-operative opioid doses are determined based on various patient factors such as pre-operative opioid use, patient weight, age and sensitivity to opioids during surgery. Patients' requirements may be underestimated and opioid regimens need to be escalated in the first 24 hours in order to alleviate uncontrolled pain in cannabis users. Better understanding of the impacts of cannabis use on post-operative opioid requirements would help the Acute Pain Service optimize post-operative pain management for patients who use cannabis pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate and signed consent form.
2. Age: 18-65 years.
3. Elective IBD bowel surgery under general anesthesia.
4. PCA use.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Elective IBD bowel surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 2 years
  Amount of morphine equivalents on PCA

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai Health System, Toronto, Ontario, Canada